CLINICAL TRIAL: NCT03646175
Title: Acute Choline Supplementation and Cardiovascular Health in Adults
Brief Title: Choline Supplementation and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Kevin Davy, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 17-562
Record Dates: First submitted 2018-08-18; First posted 2018-08-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Risk Factor
Keywords: Choline; Trimethylamine N-Oxide; Vascular health
MeSH Terms: interventions — Choline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Choline Supplementation (Experimental): Participants will consume 1000 mg (2x500 mg) of choline bitartrate the evening before each testing session.
  Interventions: Dietary Supplement: Choline
- Placebo Supplementation (Placebo Comparator): Participants will consume 1000 mg (2x500 mg) of placebo the evening before each testing session.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Choline — Participants will consume 1000 mg (2x500 mg) of choline bitartrate (over-the-counter supplement) between 10PM and 12AM the evening before the scheduled testing session and arrive fasted to the laboratory. There will be 2 testing sessions separated by 1 week.
  Arms: Acute Choline Supplementation
Dietary Supplement: Placebo — Participants will consume 1000 mg (2x500 mg) of placebo between 10PM and 12AM the evening before the scheduled testing session and arrive fasted to the laboratory. There will be 2 testing sessions separated by 1 week.
  Arms: Placebo Supplementation

SUMMARY:
Trimethylamine-N-oxide (TMAO), a metabolite produced by gut microbial metabolism of dietary choline, has recently been causally linked to atherosclerosis in animal models and has been shown to be predictive of cardiovascular disease (CVD) risk in some but not all cohort studies. The relevance of observations in animals to humans is unclear and little information is available on the mechanisms linking TMAO to increased CVD risk. Vascular dysfunction plays a critical role in the initiation and progression of atherothrombotic disease. Whether TMAO impairs vascular function in humans is not known. The purpose of this study is to determine if acute supplementation of dietary choline, which increases TMAO, impairs vascular function.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Healthy
* Non-smoking
* Weight stable for previous 6 months (±2.0 kg)
* BMI <35 kg/m^2
* Verbal and written informed consent
* Approved for participation by study medical director (Jose Rivero, M.D.)

Exclusion Criteria:

* Smoking
* Pregnancy
* Obese (BMI>35 kg/m2)
* Altered dietary patterns within the last month of recruitment
* Unstable heart disease or diabetes
* Untreated high blood pressure or high cholesterol
* Allergies to choline
* Unvaccinated against COVID-19

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Change in brachial artery function after supplementation | 30-minute measurement in laboratory
  Brachial artery function or flow mediated dilation (FMD), the blood flow and diameter of the brachial artery in the forearm (fMD), will be measured using a duplex ultrasound machine before and after the inflation of a blood pressure cuff on the forearm for 5 minutes and after placing a nitroglycerine tablet (0.4 mg) under the participant's tongue. This test will be conducted two times separated by about 1 week. The participant will be randomly-assigned to a supplement (choline or placebo) followed by a 1-week washout period (crossover design). The supplement will be taken with water between 10PM and 12AM the evening before the scheduled testing session. Off-line analysis of baseline and post-reactive hyperemic diameters and velocities will be performed using edge detection software (Vascular Analysis Tools, Medical Imaging Applications, Inc.).

SECONDARY OUTCOMES:
Change in arterial stiffness after supplementation | 45-minute measurement in laboratory
  The blood flow and diameter in the common arteries in the neck will be measured from the image obtained from an ultrasound unit (GE Vivid S6) equipped with a high resolution linear array transducer. For applanation tonometry, the carotid, brachial, radial and femoral artery pressure waveform and amplitude will be obtained by a fingertip probe incorporating a high-fidelity strain gauge transducer. Each of these measures are used to calculate arterial stiffness. These tests will be conducted two times separated by about 1 week. The participant will be randomly-assigned to a supplement (choline or placebo) followed by a 1-week washout period (crossover design). The supplement will be taken with water between 10PM and 12AM the evening before the scheduled testing session.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Davy, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic and State University, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No